CLINICAL TRIAL: NCT07341373
Title: A Single Bolus, 12-hour Euglycemic Clamp Study of the Safety, Pharmacokinetics (PK) and Glucodynamics (GD) of Intraperitoneal (IP) Portal Insulin U-500
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Portal Diabetes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PDI-PIU500-C001
Record Dates: First submitted 2025-11-25; First posted 2026-01-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Insulin; Intraperitoneal; Euglycemic Clamp; Diabetes Mellitus; Human Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This study will be conducted in 2 parts. Part A will comprise of a three-way crossover, single ascending doses (SAD) of 3 different dose levels of PI-U500 using a euglycemic clamp.
  Part B will comprise of a randomized, open-label, two-way and three-way crossover comparative single dose assessment of PI-U500 versus Humulin® R U-500 administered IP versus Lyumjev® U-100 subcutaneously (SC) using a euglycemic clamp.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A, Group 1, Single Ascending Dose (Experimental): Participants will receive PI-U500 intraperitoneally at 0.1 U/kg, then 0.2 U/kg and lastly 0.3 U/kg
  Interventions: Drug: Portal Insulin U-500
- Part B, Group 2 (Other): A three-way crossover where participants will receive 0.1 U/kg of PI-U500, followed by 0.2 U/kg of Humulin R U500 (Active Control), and finally 0.2 U/kg of PI-U500. All administered intraperitoneally.
  Interventions: Drug: Portal Insulin U-500; Drug: Humulin R U-500
- Part B, Group 3 (Other): A three-way crossover where participants will receive 0.1 U/kg of PI-U500, followed by 0.2 U/kg of Humulin R U500 (Active Control), and finally 0.3 U/kg of PI-U500. All administered intraperitoneally.
  Interventions: Drug: Portal Insulin U-500; Drug: Humulin R U-500
- Part B, Group 4 (Other): A three-way crossover where participants will receive 0.2 U/kg of Lyumjev U-100 (Active Control) subcutaneously, followed by 0.2 U/kg of PI-U500 intraperitoneally, and finally 0.3 U/kg of PI-U500, also intraperitoneally.
  Interventions: Drug: Portal Insulin U-500; Drug: Lyumjev U-100 Insulin
- Part B, Group 5 (Other): A two-way crossover where participants will receive 0.2 U/kg of Lyumjev U-100 (Active Control) subcutaneously, followed by 0.2 U/kg of PI-U500 intraperitoneally.
  Interventions: Drug: Portal Insulin U-500; Drug: Lyumjev U-100 Insulin
- Part B, Group 6 (Other): A three-way crossover where participants will receive 0.2 U/kg of each of the drugs sequentially, but the order will be randomized into three options:
  * Option 1: 0.2 U/kg of Lyumjev U-100 (Active Control) subcutaneously, followed by 0.2 U/kg of Humulin R U500 (Active Control) intraperitoneally, and finally 0.2 U/kg of PI-U500 intraperitoneally.
  * Option 2: 0.2 U/kg of Humulin R U500 (Active Control) intraperitoneally , followed by 0.2 U/kg of PI-U500 intraperitoneally, and finally 0.2 U/kg of Lyumjev U-100 (Active Control) subcutaneously.
  * Option 3: 0.2 U/kg of PI-U500 intraperitoneally , followed by 0.2 U/kg of Lyumjev U-100 (Active Control) subcutaneously, and finally 0.2 U/kg of Humulin R U500 (Active Control) intraperitoneally.
  Interventions: Drug: Portal Insulin U-500; Drug: Humulin R U-500; Drug: Lyumjev U-100 Insulin

INTERVENTIONS:
Drug: Portal Insulin U-500 — Intraperitoneal delivery of a single dose at 0.1 U/kg during an euglycemic clamp
  Other Names: PI-U500
  Arms: Part A, Group 1, Single Ascending Dose; Part B, Group 2; Part B, Group 3
Drug: Portal Insulin U-500 — Intraperitoneal delivery of a single dose at 0.2 U/kg during an euglycemic clamp
  Other Names: PI-U500
  Arms: Part A, Group 1, Single Ascending Dose; Part B, Group 2; Part B, Group 4; Part B, Group 5; Part B, Group 6
Drug: Portal Insulin U-500 — Intraperitoneal delivery of a single dose at 0.3 U/kg during an euglycemic clamp
  Other Names: PI-U500
  Arms: Part A, Group 1, Single Ascending Dose; Part B, Group 3; Part B, Group 4
Drug: Humulin R U-500 — Intraperitoneal delivery of a single dose at 0.2 U/kg during an euglycemic clamp
  Arms: Part B, Group 2; Part B, Group 3; Part B, Group 6
Drug: Lyumjev U-100 Insulin — Subcutaneous delivery of a single dose at 0.2 U/kg during an euglycemic clamp
  Arms: Part B, Group 4; Part B, Group 5; Part B, Group 6

SUMMARY:
The goal of this clinical trial is to assess the safety of a new U500 insulin formulation and to determine how rapidly it is absorbed and how long it takes to act when administered intraperitoneally. The trial will be conducted in people with Type 1 Diabetes. The main questions it aims to answer are:

Is the drug safe and tolerable when administered intraperitoneally? How fast is it absorbed, and how long does it take to act? Researchers will compare the investigational product (PI-U500) with Humulin R U500 administered intraperitoneally and Lyumjev U100 administered subcutaneously.

Participants will undergo a 12-hour clamp procedure in which their blood glucose will be maintained stable via glucose infusion at variable rates after a single intraperitoneal injection of the insulin formulation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet all the following criteria at Screening will be included in the study:

  1. Subjects ≥18 to ≤60 years of age at the time of signing the informed consent.
  2. Subjects diagnosed with T1DM for at least 12 months.
  3. Subjects who have been using an approved insulin pump or use MDI with basal and bolus insulin (stable use for 3 months).
  4. Fasting C-peptide concentration of ≤0.3 nmol/L (0.9061 ng/ml), assessed at a plasma glucose concentration >90 mg/dL. (If necessary, the subject may consume carbohydrates to raise BG over 90 mg/dL as measured by YSI (glucose analyzer) prior to drawing blood for C-peptide. This may be repeated as needed to ensure C-peptide is assessed when plasma glucose concentration is >90 mg/dL).
  5. HbA1c concentration of ≤8.5%.
  6. Body mass index (BMI) within the range ≥18.5 to ≤30.0 kg/m2.
  7. Weight ≥ 50 kg.
  8. Female subjects must be non-pregnant and non-lactating and postmenopausal (no menses >12 months); postmenopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels at Screening for all female subjects.
  9. Male subjects must be surgically sterile, abstinent or if engaged in sexual relations of child-bearing potential, the subject and his partner must be using acceptable methods of contraception.
  10. Has venous access sufficient to allow for blood sampling.
  11. Capable of giving signed informed consent and willing to follow study procedures and commitment to the study duration.

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from participating in the study:

  1. A subject who has proliferative retinopathy or maculopathy (based on records/documentation of ophthalmologic exam within 18 months of Screening or ophthalmologic exam during Screening), severe gastroparesis, and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator.
  2. History of ≥2 episodes of severe hypoglycemia (as defined per ADA criteria) or ≥1 episodes of diabetic ketoacidosis or emergency room visits for uncontrolled diabetes leading to hospitalization within 6 months prior to Screening.
  3. Subject is not able to avoid major dietary changes for the duration of the study.
  4. Systolic blood pressure >150 mm Hg and/or diastolic blood pressure >90 mm Hg at Screening. Treatment with no more than 2 antihypertensive medications must be with stable doses for at least 3 months prior to Screening.
  5. Current use of any drugs as listed in the table of prohibited medications.
  6. History of any major surgery within 6 months prior to Screening.
  7. History of any serious allergic adverse reaction or hypersensitivity to any of the product components.
  8. History of renal disease or abnormal kidney function tests at Screening (GFR <60 mL/min/1.73m2 as estimated using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]).
  9. Triglycerides >500 mg/dL at Screening.
  10. Clinically significant abnormal hematology or biochemistry screening tests. Subjects may have these labs be redrawn once on a separate day.
  11. Any history of heart disease, defined as symptomatic heart failure (New York Heart Association class III or IV), myocardial infarction, coronary artery bypass graft surgery, or angioplasty, unstable angina requiring medication, transient ischemic attack, cerebral infarct, or cerebral hemorrhage.
  12. Presence of clinically significant physical, laboratory, or ECG findings (eg, QTcF >450 msec for males, QTcF >470 msec for females) at Screening that, in the opinion of the Investigator, may interfere with any aspect of study conduct or interpretation of results.
  13. History or presence of malignant neoplasms within the past 5 years prior to the day of Screening. Basal and squamous cell skin cancer and any in-situ carcinomas are allowed.
  14. Clinically significant concomitant disease including cardiovascular, renal, hepatic, respiratory, gastrointestinal, hematological, dermatological, neurological, psychiatric, systemic or infections disease as judged by the Investigator.
  15. Personal or family history of hypercoagulability or thromboembolic disease.
  16. History of any active infection, other than mild viral illness within 30 days prior to dosing as judged by the Investigator.
  17. Administration of any vaccinations in the 2 weeks prior to admission to the clinic.
  18. History of alcohol abuse as judged by the Investigator within approximately 1 year or consuming >2 standard drinks on average per day in men, and >1 standard drinks on average per day in women, and/or positive alcohol breath test at Screening or upon clinic admission. (One drink is defined as 12 fluid ounces of regular beer [5% alcohol], 5 fluid ounces of wine [12% alcohol], or 1.5 fluid ounces of 80 proof [40% alcohol] distilled spirits.)
  19. History of illicit/recreational drug abuse within approximately 1 year as judged by the Investigator. Frequent use of marijuana or other tetrahydrocannabinol (THC) products within 6 weeks, or clinically under the effect at Screening or upon clinic admission, as per Investigator evaluation or a positive urine drug test at Screening or upon clinic admission.
  20. Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day); or non- or occasional smoker who is not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period.
  21. Known history or positive test of hepatitis B surface antigen (HBsAg), hepatitis C antibody test (anti-HCV), or human immunodeficiency virus type 1 (HIV-1) or 2 (HIV-2) antibody at Screening.
  22. Existence of any surgical or medical condition that, in the judgment of the Investigator, might interfere with the absorption, distribution or metabolism of the drugs or the tolerability/safety measurements.
  23. Any subject who, per the opinion of the Investigator, will not make a good study subject relative to mental disorder, history of poor treatment adherence, etc.
  24. Participation in an investigational study within 30 days prior to dosing or within 5 half-lives of the last dose of study drug whichever is longer.
  25. Donation or loss of >500 mL of blood or blood product within 56 days of Screening.
  26. Poor venous access as judged by the study team.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | From enrollment until the follow-up visit, an average of 2 months
Safety: Change from baseline in systolic and diastolic blood pressure | Will be measured at 2 times, first within 4 hours before drug administration (Pre-clamp) and then after 12 hours of drug administration (post-clamp)
Safety: Change from baseline in temperature | Will be measured at 2 times, first within 4 hours before drug administration (Pre-clamp) and then after 12 hours of drug administration (post-clamp)
Safety: Change from baseline in respiratory rate | Will be measured at 2 times, first within 4 hours before drug administration (Pre-clamp) and then after 12 hours of drug administration (post-clamp)
Safety: Change from baseline in heart rate | Will be measured at 2 times, first within 4 hours before drug administration (Pre-clamp) and then after 12 hours of drug administration (post-clamp)
Safety: Change from baseline in 12-lead electrocardiogram (ECG) parameters | Pre-dose and after the end of PK-sampling (720 minutes post-dose)
  The following parameters will be recorded from the subject's ECG trace as calculated by the machine algorithm: heart rate, QT interval, PR interval, QRS interval, RR interval, and QTc (corrected) using the Fridericia correction (QTcF = QT ÷ cube root of the R-R interval [where R-R is the duration of the entire cardiac cycle]).
Safety: Incidence and severity of clinical findings on physical examination | Pre-dose and after the end of PK-sampling (720 minutes post-dose)
Tolerability: Pain assessments per Visual Analogue Scale (VAS) | 10 min and 1 hour post-dosing
  VAS assessment will target the assessment of abdominal pain. The scale will go from 0 to 10, with 10 being the maximum pain.
Tolerability: Change in Interleukin 6 [IL-6] levels | Blood samples will be taken immediately before dosing, 2 hours after dosing, and with the last PK sample (720 minutes after dosing)
Tolerability: Change in tumor necrosis factor [TNF-α] levels | Blood samples will be taken immediately before dosing, 2 hours after dosing, and with the last PK sample (720 minutes after dosing)
Tolerability: Change in high sensitivity C-reactive protein [hsCRP] levels | Blood samples will be taken immediately before dosing, 2 hours after dosing, and with the last PK sample (720 minutes after dosing)
Pharmacokinetic: Area under the insulin concentration-time curve (AUC) | From the time of dose (time 0) until 12 hours post-dose (AUCIns,0-12h)
  For the duration of the euglycemic clamp
Pharmacokinetic: Maximum insulin concentration (Cmax) | Over 12 hours post-dosing
Pharmacokinetic: Time to maximum insulin concentration (Tmax) | Over 12 hours post-dosing
Glucodynamic: Area under the glucose infusion rate (GIR) time curve | From the time of dose (time 0) until 12 hours post-dose (AUCGIR,0-12h)
Glucodynamic: Maximum GIR (GIRmax) | Over 12 hours post-dosing
Glucodynamic: Time to maximum GIR (TGIRmax) | Over 12 hours post-dosing

SECONDARY OUTCOMES:
Pharmacokinetic: Area under the partial insulin concentration-time curves (AUC) in time intervals | From 0 to 15 minutes (AUCIns,0-15 min), from 0-30 minutes (AUCIns,0-30 min) and from 3 hours to end (AUCIns,3h-end)
Pharmacokinetic: Time to half-maximum insulin concentration before Cmax (t50%-INS (early)) | Over 12 hour post-dosing
Pharmacokinetic: Time to half-maximum insulin concentration after Cmax (t50%-INS (late)) | Over 12 hours post-dosing
Pharmacokinetic: Onset of appearance | Over 12 hours post-dosing
  Defined as time from study drug administration until the first time insulin concentrations were equal to or higher than the lower limit of quantification
Glucodynamic: Area under GIR time curve in time intervals | From 0-30 minutes (AUCGIR,0-30 min), from 0 to 1 hour (AUCGIR,0-1h), from 4 hours to end (AUCGIR,4h-end), from 0 to 6 hours (AUCGIR,0-6h) and from 0 to end (AUCGIR,0-end)
Glucodynamic: Time to half-maximum GIR before GIRmax (t50%-GIR (early)) | Over 12 hours post-dosing
Glucodynamic: Time to half-maximum GIR after GIRmax (t50%-GIR (late)) | Over 12 hours post-dosing

CONTACTS AND LOCATIONS:
Locations (1):
- ProSciento, Inc., Chula Vista, California, United States